CLINICAL TRIAL: NCT03613740
Title: Effect of Fucoxanthin on the Metabolic Syndrome, Insulin Sensitivity and Insulin Secretion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Karina Griselda Pérez Rubio, Principal Investigator, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fucoxanthin-MS
Record Dates: First submitted 2018-07-19; First posted 2018-08-03 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-09

CONDITIONS: Metabolic Syndrome
Keywords: Insulin Sensitivity; Metabolic Syndrome; Fucoxanthin; Insulin Secretion
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance | interventions — fucoxanthin; stearic acid

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fucoxanthin (Experimental): 12 mg Fucoxanthin capsule, once a day before breakfast during 90 days.
  Interventions: Drug: Fucoxanthin
- Placebo (Placebo Comparator): Homologated magnesium sterate capsule, once a day before breakfast during 90 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fucoxanthin — Intervention will be administered 30 minutes before breakfast.
  Arms: Fucoxanthin
Drug: Placebo — Intervention will be administered 30 minutes before breakfast.
  Other Names: Magnesium Sterate
  Arms: Placebo

SUMMARY:
The Metabolic Syndrome (MS) is a cluster of cardiometabolic risk factors, which include abdominal obesity, hyperglycemia, dyslipidemia, and high blood pressure. MS is considered a serious problem to health systems due to a current inability on implementing an effective prevention and treatment program. In Mexico 73% of adult population suffers obesity or overweight, this condition triggers the best studied pathophysiological mechanism; insulin resistance, which in turn precedes the diagnosis of diabetes and cardiovascular disease, that are the main cause of general mortality in Mexico, thus the prevention and timely treatment of this condition are now a priority.

Actual pharmacological therapy is designed to control its components individually, however, there are great interest in developing new therapeutic lines that improve more than one component simultaneously and thereby increase the cost-benefit and effectiveness of the therapy. Fucoxanthin is a functional element present in seaweed species. Several studies have offered certain perspectives on its action mechanism and safety. The information available is favorable for weight control in overweight subjects, but its activity in glucose levels, lipid metabolism and blood pressure is inconsistent. It represents a natural option with great interest in this research, since it could be a new, safe and effective therapy in the MS.

The aim of this study is to evaluate the effect of fucoxanthin on the components of the MS, insulin sensitivity and insulin secretion. The investigators hypothesis is that Fucoxanthin modifies the components of the MS, insulin sensitivity and insulin secretion

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, clinical trial will be conducted in 28 patients with MS according to the International Diabetes Federation (IDF) criteria, men and women, ages 30 to 60. Participants will be assigned randomly into two groups of 14 individuals each. Patients will receive a capsule with Fucoxanthin 12 mg or homologated placebo once a day during 90 days.

Waist circumference, fasting blood glucose, serum triglycerides, serum HDL cholesterol and blood pressure will be evaluated before and after intervention in both groups. First phase of insulin secretion (Stumvoll index), total insulin secretion (Insulinogenic index) and Insulin sensitivity (Matsuda index) will be calculated from the concentration of glucose and insulin obtained from an Oral Glucose Tolerance Test.

Data from statistical analysis will be presented through measures of central tendency and dispersion( mean and standard deviation) for quantitative variables and frequencies and percentages for qualitative variables. The qualitative variables will be analyzed through the X2 or Fisher's exact test. The intra-group analysis of the quantitative variables will be carried out by means of the Wilcoxon rank test, while the inter-group analysis with the U test of Mann Whitney and Kruskal-Wallis. Statistical significance will be considered with a p<0.05.

This protocol was approved by a local ethics committee and written informed consent will be obtained from all volunteers

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed MS according to the IDF criteria:
* - - Waist circumference: ≥80 cm (women) ≥90 cm (men), plus two or more of the following:
* - - - - Fasting glucose ≥ 100 mg/dL
* - - - - Triglycerides ≥150 mg/dL
* - - - - HDL-C: Men ≤40 mg/dL, women ≤50 mg/dL
* - - - - Blood pressure ≥130/85 mmHg
* Body Mass Index between 25 and 34.9 kg/m²
* No pharmacological treatment for MS
* Stable weight during the last 3 months

Exclusion Criteria:

* Pregnancy or breast-feeding
* History of kidney or liver disease
* Drugs or supplements consumption with proven properties that modify the behavior of the MS
* Total cholesterol >240 mg/dL
* Triglycerides >500mg/dL
* Glucose ≥126 mg/dL or HbA1C ≥6.5%.
* Hypersensitivity to Fucoxanthin

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Gonzalez Ortiz, MD MSc Phd, Principal Investigator — University of Guadalajara
Locations (1):
- Instituto de Terapeútica Experimental y Clínica. Centro Universitario de Ciencias de la Salud. Universidad de Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lopez-Ramos A, Gonzalez-Ortiz M, Martinez-Abundis E, Perez-Rubio KG. Effect of Fucoxanthin on Metabolic Syndrome, Insulin Sensitivity, and Insulin Secretion. J Med Food. 2023 Jul;26(7):521-527. doi: 10.1089/jmf.2022.0103. Epub 2023 Jul 4. PMID 37405785
- [Derived] Yang M, Xuan Z, Wang Q, Yan S, Zhou D, Naman CB, Zhang J, He S, Yan X, Cui W. Fucoxanthin has potential for therapeutic efficacy in neurodegenerative disorders by acting on multiple targets. Nutr Neurosci. 2022 Oct;25(10):2167-2180. doi: 10.1080/1028415X.2021.1926140. Epub 2021 May 15. PMID 33993853

RESULTS

PARTICIPANT FLOW:
Groups:
- Fucoxanthin: Received one (1) 12 mg fucoxanthin capsule, once a day.
- Placebo: Received one (1) Magnesium stearate capsule, once a day
Period: Overall Study
Arm/Group | Fucoxanthin | Placebo
Started | 14 | 14
Completed | 13 | 13
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fucoxanthin | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (7.8) | 45.6 (9.1) | 47.4 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 7 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 14 | 28
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 14 | 14 | 28
Waist Circumference [Mean (Standard Deviation); unit: cm] | 101.2 (9.1) | 102.1 (5.0) | 101.7 (7.2)
Body Weight [Mean (Standard Deviation); unit: kg] | 80.6 (11.2) | 80.9 (8.6) | 80.7 (9.8)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.1 (3.6) | 30.7 (2.3) | 30.9 (3.0)
Body Fat [Mean (Standard Deviation); unit: Percentage] | 34.6 (8.6) | 34.3 (6.8) | 34.4 (7.6)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 126.1 (10.3) | 120.8 (15.7) | 124.1 (13.3)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 81.5 (6.5) | 80.3 (8.8) | 80.9 (7.6)
Fasting Serum Glucose [Mean (Standard Deviation); unit: mmol/L] | 5.5 (0.6) | 5.7 (0.5) | 5.6 (0.5)
Triglycerides [Mean (Standard Deviation); unit: mmol/L] | 2.2 (0.7) | 2.4 (1.0) | 2.3 (0.9)
Total Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 5.3 (1.0) | 5.0 (0.9) | 5.1 (1.0)
High-Density Lipoprotein (HDL-C) [Mean (Standard Deviation); unit: mmol/L] | 1.2 (0.3) | 1.2 (0.2) | 1.2 (0.2)
Low-Density lipoprotein (LDL-C) [Mean (Standard Deviation); unit: mmol/L] | 3.1 (1.0) | 2.67 (0.9) | 2.9 (1.0)
Very-Low-Density Lipoprotein (VLDL) [Mean (Standard Deviation); unit: mmol/L] | 1.0 (0.3) | 1.1 (0.5) | 1.0 (0.5)
Matsuda-DeFronzo insulin sensitivity index [Mean (Standard Deviation); unit: Index] — The Matsuda-DeFronzo index measures whole-body insulin sensitivity from serum insulin and glucose levels during an oral glucose tolerance test (OGTT). The index is calculated with the formula: 10,000 / sqrt([fasting glucose (mg/dL) × fasting insulin (µU/mL)] × [mean glucose × mean insulin during OGTT]). The scale ranges from 0 to infinity, with higher values indicating greater insulin sensitivity. Typical values for healthy individuals range between 2 and 10, while lower values suggest insulin resistance.
  Index | 2.07 (0.74) | 2.12 (1.10) | 2.10 (0.92)
Stumvoll index [Mean (Standard Deviation); unit: Index] — The Stumvoll index measures the first phase of insulin secretion, incorporates demographic data along with plasma glucose (mmol/L) and insulin (pmol/L) levels measured during an oral glucose tolerance test (OGTT). There is no universally standardized ranges, values ranges from 0 to infinity; higher values indicate a better early insulin response to glucose (first 30 minutes), reflecting more effective beta-cell function.
  Index | 2403 (621) | 2155 (698) | 2279 (660)
Total Insulin Secretion [Mean (Standard Deviation); unit: Ratio] — The Total Insulin Secretion is calculated as the ratio of the area under the curve (AUC) for insulin to the AUC for glucose during a 120-minute oral glucose tolerance test (OGTT). The formula is: AUC insulin / AUC glucose. AUC values are derived from concentrations measured at 0, 30, 60, 90, and 120 minutes post-ingestion of a glucose solution at baseline day. Interpretation of the AUC insulin/AUC glucose ratio is as follows: values <0.5 indicate insulin resistance, values between 0.5 and 1.0 suggest moderate insulin secretion, and values >1.0 reflect optimal insulin secretion.
  Ratio | 0.84 (0.31) | 0.80 (0.21) | 0.82 (0.27)
Alanine Aminotransferase [Mean (Standard Deviation); unit: ukat/L] | 0.45 (0.29) | 0.53 (0.32) | 0.49 (0.30)
Aspartate Aminotransferase [Mean (Standard Deviation); unit: ukat/L] | 0.39 (0.31) | 0.40 (0.26) | 0.40 (0.28)
Creatinin [Mean (Standard Deviation); unit: µmol/L] | 78.4 (23.6) | 86.9 (32.6) | 82.6 (28.3)

OUTCOME MEASURES:

1. Primary Outcome: Waist Circumference (WC)
Description: WC was measured with a flexible tape at the midline between the highest point of the iliac crest and the lowest rib in the midaxillary line.
Time Frame: 12 weeks.
Population: All participants, including those who dropped out before the end were taken into account for statistical analysis (intention to treat)
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Fucoxanthin | Placebo
Number analyzed (Participants) | 13 | 13
cm | 98.9 (9.3) | 102.1 (5.6)

2. Primary Outcome: Fasting Serum Glucose
Description: Fasting serum glucose concentration was measured with enzymatic/colorimetric techniques by spectrophotometry.
Time Frame: 12 weeks.
Population: All participants, including those who dropped out before the end of the study were taken into account for statistical analysis (intention to treat)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Fucoxanthin | Placebo
Number analyzed (Participants) | 13 | 13
mmol/L | 5.5 (0.6) | 5.6 (0.5)

3. Primary Outcome: Triglycerides (TG)
Description: TG concentration was measured with enzymatic/colorimetric techniques by spectrophotometry.
Time Frame: 12 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Fucoxanthin | Placebo
Number analyzed (Participants) | 13 | 13
mmol/L | 2.1 (0.7) | 2.4 (0.9)

4. Primary Outcome: High-Density Lipoprotein (HDL-C)
Description: Serum HDL-C concentration was measured with enzymatic/colorimetric techniques by spectrophotometry.
Time Frame: 12 weeks.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Fucoxanthin | Placebo
Number analyzed (Participants) | 13 | 13
mmol/L | 1.2 (0.2) | 1.2 (0.2)

5. Primary Outcome: Systolic Blood Pressure
Description: Blood pressure was evaluated using a digital sphygmomanometer after a resting period of 15 min with the subject sitting; the bracelet was adjusted 3.0 cm above the fold of the elbow of the left arm.
Time Frame: 12 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Fucoxanthin | Placebo
Number analyzed (Participants) | 13 | 13
mmHg | 120.8 (9.7) | 119.1 (14.5)

6. Primary Outcome: Diastolic Blood Pressure
Description: as for outcome 5
Time Frame: 12 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Fucoxanthin | Placebo
Number analyzed (Participants) | 13 | 13
mmHg | 78.6 (6.3) | 79.2 (7.4)

7. Primary Outcome: Matsuda-DeFronzo Insulin Sensitivity Index
Description: The Matsuda-DeFronzo index measures whole-body insulin sensitivity from serum insulin and glucose levels during an oral glucose tolerance test (OGTT). The index is calculated with the formula: 10,000 / sqrt([fasting glucose (mg/dL) × fasting insulin (µU/mL)] × [mean glucose × mean insulin during OGTT]). The scale ranges from 0 to infinity, with higher values indicating greater insulin sensitivity. Typical values for healthy individuals range between 2 and 10, while lower values suggest insulin resistance.
Time Frame: 12 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Fucoxanthin | Placebo
Number analyzed (Participants) | 13 | 13
index | 2.19 (0.90) | 2.19 (1.07)

8. Primary Outcome: Total Insulin Secretion
Description: The Total Insulin Secretion is calculated as the ratio of the area under the curve (AUC) for insulin to the AUC for glucose during a 120-minute oral glucose tolerance test (OGTT). The formula is: AUC insulin / AUC glucose. AUC values are derived from concentrations measured at 0, 30, 60, 90, and 120 minutes post-ingestion of a glucose solution at week 12. Interpretation of the AUC insulin/AUC glucose ratio is as follows: values <0.5 indicate insulin resistance, values between 0.5 and 1.0 suggest moderate insulin secretion, and values >1.0 reflect optimal insulin secretion.
Time Frame: 12 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Fucoxanthin | Placebo
Number analyzed (Participants) | 13 | 13
Ratio | 1.02 (0.32) | 0.85 (0.23)

9. Primary Outcome: Stumvoll Index
Description: The Stumvoll index measures the first phase of insulin secretion, incorporates demographic data along with plasma glucose (mmol/L) and insulin (pmol/L) levels measured during an oral glucose tolerance test (OGTT). There is no universally standardized ranges, values ranges from 0 to infinity; higher values indicate a better early insulin response to glucose (first 30 minutes), reflecting more effective beta-cell function.
Time Frame: 12 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Fucoxanthin | Placebo
Number analyzed (Participants) | 13 | 13
index | 2907 (732) | 2298 (446)

10. Secondary Outcome: Body Weight
Description: Body weight was measured at baseline a bioimpedance scale.
Time Frame: 12 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Fucoxanthin | Placebo
Number analyzed (Participants) | 13 | 13
kg | 79.16 (12.3) | 82.1 (7.9)

11. Secondary Outcome: Body Mass Index (BMI)
Description: BMI was calculated with the Quetelet index formula.
Time Frame: 12 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Fucoxanthin | Placebo
Number analyzed (Participants) | 13 | 13
kg/m^2 | 30.3 (3.7) | 31.0 (2.1)

12. Secondary Outcome: Body Fat
Description: Percentage of body fat was measured using a bioimpedance scale.
Time Frame: 12 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Fucoxanthin | Placebo
Number analyzed (Participants) | 13 | 13
percentage | 33.0 (8.3) | 34.9 (7.4)

13. Secondary Outcome: Total Cholesterol (TC)
Description: Serum Total Cholesterol concentration was measured with enzymatic/colorimetric techniques by spectrophotometry.
Time Frame: 12 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Fucoxanthin | Placebo
Number analyzed (Participants) | 13 | 13
mmol/L | 5.1 (1.0) | 4.9 (1.0)

14. Secondary Outcome: Low-Density Lipoprotein (LDL-C)
Description: Serum LDL-C concentration was calculated using the Friedewald formula (LDL-C = TC - (HDL-C + [TG/5])
Time Frame: 12 weeks.
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Fucoxanthin | Placebo
Number analyzed (Participants) | 13 | 13
mmol/L | 3.0 (0.9) | 2.7 (1.0)

15. Secondary Outcome: Very-Low-Density Lipoprotein (VLDL)
Description: Serum VLDL concentration was calculated with the formula: VLDL-C = TG/5.
Time Frame: 12 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Fucoxanthin | Placebo
Number analyzed (Participants) | 13 | 13
mmol/L | 0.9 (0.3) | 1.1 (0.4)

16. Secondary Outcome: Alanine Aminotransferase (ALT)
Description: Serum ALT concentration was measured with enzymatic/colorimetric techniques by spectrophotometry.
Time Frame: 12 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ukat/L
Arm/Group | Fucoxanthin | Placebo
Number analyzed (Participants) | 13 | 13
ukat/L | 0.47 (0.24) | 0.50 (0.29)

17. Secondary Outcome: Aspartate Aminotransferase (AST)
Description: Serum AST concentration was measured with enzymatic/colorimetric techniques by spectrophotometry.
Time Frame: 12 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ukat/L
Arm/Group | Fucoxanthin | Placebo
Number analyzed (Participants) | 13 | 13
ukat/L | 0.41 (0.28) | 0.42 (0.26)

18. Secondary Outcome: Creatinin
Description: Serum creatinin concentration was measured with enzymatic/colorimetric techniques by spectrophotometry.
Time Frame: 12 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Fucoxanthin | Placebo
Number analyzed (Participants) | 13 | 13
µmol/L | 83.8 (21.7) | 76.4 (26.4)

ADVERSE EVENTS:
Time Frame: 12 weeks.
Description: Adverse event and serious adverse event definition does not differ from the clinicaltrials.gov definitions.
Arm/Group | Fucoxanthin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 5/14 | 5/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fucoxanthin (N=14) | Placebo (N=14)
Frequent bowel movements (Gastrointestinal disorders) | 4 (4) | 3 (3)
Flatulence (Gastrointestinal disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT03613740/Prot_SAP_ICF_000.pdf